CLINICAL TRIAL: NCT01516710
Title: Prospective Randomized Study of Laparoscopic Versus Open Liver Resection for Colorectal Metastases
Brief Title: Oslo Randomized Laparoscopic Versus Open Liver Resection for Colorectal Metastases Study
Acronym: Oslo-CoMet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Åsmund Avdem Fretland, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/1285/REK sør-øst B
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-11

CONDITIONS: Secondary Malignant Neoplasm of Liver; Colorectal Neoplasms
Keywords: Open liver resection; Laparoscopic liver resection; Colorectal cancer liver metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open liver resection (Active Comparator): Patients will be operated with open liver resection
  Interventions: Procedure: Open liver resection
- Laparoscopic liver resection (Active Comparator): Patients will be operated with laparoscopic liver resection
  Interventions: Procedure: Laparoscopic liver resection

INTERVENTIONS:
Procedure: Open liver resection — Patients will be operated with open liver resection for colorectal metastasis
  Other Names: Open liver resection using standard technique:; Ligasure; CUSA; Thunderbeat; Autosonix; SonoSurg; Ultrasound
  Arms: Open liver resection
Procedure: Laparoscopic liver resection — Patients will be operated with laparoscopic liver resection
  Other Names: Laparoscopic liver resection using standardized technique:; Ligasure; CUSA; Thunderbeat; Autosonix; SonoSurg; Laparoscopic ultrasound
  Arms: Laparoscopic liver resection

SUMMARY:
The purpose of the study is to compare outcomes of laparoscopic versus open liver resection for colorectal metastases in a prospective and randomized study. The study will include all non-anatomic liver resections in our institution.

The primary end point is that the use of laparoscopic technique significantly can reduce the frequency of complications to liver resection. Secondary end points are 5-year survival, immediate surgical outcomes, quality of life and degree of impairment of the immune system.

DETAILED DESCRIPTION:
Full protocol is published open access in Trialsjournal:

http://www.trialsjournal.com/content/16/1/73

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for radical liver resection without formal liver resection or without assistance of radiofrequency ablation

Exclusion Criteria:

* Inability to give written informed concent
* Patients with tumors that can't be resected without reconstruction of vessels or bile ducts
* Patients with tumors that can't be resected without 1)formal liver resection 2)combination with radiofrequency ablation
* Patients with extrahepatic metastasis except resectable metastasis in lungs and adrenals
* Pre- and peroperative diagnosis of non radically treatable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Edwin, MD, PhD, Study Chair — Oslo University Hospital - The Interventional Centre; Bjorn Edwin, MD, PhD, Principal Investigator — Oslo University Hospital - The Interventional Centre
Locations (1):
- Oslo University Hospital, Department of Gastrointestinal surgery, The National Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Not decided yet but results will be public no matter the outcome of the trial

REFERENCES:
- [Derived] Aghayan DL, Kazaryan AM, Dagenborg VJ, Rosok BI, Fagerland MW, Waaler Bjornelv GM, Kristiansen R, Flatmark K, Fretland AA, Edwin B; OSLO-COMET Survival Study Collaborators. Long-Term Oncologic Outcomes After Laparoscopic Versus Open Resection for Colorectal Liver Metastases : A Randomized Trial. Ann Intern Med. 2021 Feb;174(2):175-182. doi: 10.7326/M20-4011. Epub 2020 Nov 17. PMID 33197213
- [Derived] Fretland AA, Dagenborg VJ, Waaler Bjornelv GM, Aghayan DL, Kazaryan AM, Barkhatov L, Kristiansen R, Fagerland MW, Edwin B, Andersen MH. Quality of life from a randomized trial of laparoscopic or open liver resection for colorectal liver metastases. Br J Surg. 2019 Sep;106(10):1372-1380. doi: 10.1002/bjs.11227. Epub 2019 Jul 19. PMID 31322735
- [Derived] Fretland AA, Kazaryan AM, Bjornbeth BA, Flatmark K, Andersen MH, Tonnessen TI, Bjornelv GM, Fagerland MW, Kristiansen R, Oyri K, Edwin B. Open versus laparoscopic liver resection for colorectal liver metastases (the Oslo-CoMet Study): study protocol for a randomized controlled trial. Trials. 2015 Mar 4;16:73. doi: 10.1186/s13063-015-0577-5. PMID 25872027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Liver Resection | Laparoscopic Liver Resection
Started | 147 | 133
Completed | 143 | 129
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: A total of 280 patients were enrolled. Only 273 underwent surgery, and only these could reach the primary endpoint of 30 days morbidity. This is why there is a difference between baseline and analyzed for the primary endpoint.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Liver Resection | Laparoscopic Liver Resection | Total
Number analyzed (Participants) | 147 | 133 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 67 (8) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 56 | 116
  Male | 87 | 77 | 164
Region of Enrollment [Count of Participants; unit: Participants] — Region of enrollment is Norway
  Participants
    Norway | 147 | 133 | 280

OUTCOME MEASURES:

1. Primary Outcome: 30 Days Perioperative Morbidity
Description: This study aims to compare major intraoperative and postoperative parameters in patients randomized to either laparoscopic or open liver resection. Pre- and perioperative events relevant for surgical outcomes will be registered. The following intraoperative parameters will be compared: operative time, blood loss, blood transfusion, while intraoperative incidents will be classified according to the Satava classification. Morbidity within the first 30 days is the primary outcome (morbidity, yes/no), and will be classified and analysed according to the validated classification for postoperative morbidity as described by Dindo et al, by the Accordion system and by the Comprehensive Complication Index
Time Frame: Within 30 days after surgery
Population: Modified intention to treat
Measure: Number; unit: Complications Accordion grade 2 or highe
Arm/Group | Open Liver Resection | Laparoscopic Liver Resection
Number analyzed (Participants) | 144 | 129
Complications Accordion grade 2 or highe | 44 | 24

2. Secondary Outcome: 5 Year Survival
Description: 5 year survival
  * overall
  * disease free
  * recurrence free
Time Frame: 5 years after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Recurrence Pattern
Description: Pattern of recurrence in liver and extrahepatic. Studied by postoperative CT every 4 months for 2 years and every 6 months for the following 3 years. Local recurrence and new tumors will be recorded.
Time Frame: 5 years
Reporting Status: Not Posted

4. Secondary Outcome: Immediate Oncologic Outcome
Description: Immediate oncologic outcome is the result of surgical specimen evaluation - evaluation of tumor resection margins.
Time Frame: 2 months after surgery
Reporting Status: Not Posted

5. Secondary Outcome: Postoperative Quality of Life
Description: Evaluation of postoperative quality of life at baseline, 1 month, 4 months and 2 years using the SF-36 and the EORTC qlq-30 lmc-21 forms
Time Frame: Up to 2 years
Reporting Status: Not Posted

6. Secondary Outcome: Surgical Trauma and Activation of the Immune System
Description: Evaluation of surgical trauma caused by open and laparoscopic resection by means of analyzing complement and cytokine activation at set perioperative time points.
Time Frame: 72 hours
Reporting Status: Not Posted

7. Secondary Outcome: Health Economy
Description: We intend to compare overall cost of treatment for the hospital and for the health care system
Time Frame: 1 year
Reporting Status: Not Posted

8. Secondary Outcome: Severity of Postoperative Pain
Description: To compare pain the first 5 postoperative days, at 1 month and 4 months. Patients in the open group will be randomized to receiving either a patient controlled analgesic pump containing opioids, or a patient controlled epidural analgesic pump. In laparoscopic group all patients will receive a PCA.
Time Frame: 4 months
Reporting Status: Not Posted

9. Secondary Outcome: Molecular Biology
Description: The aim is to perform molecular characterization of biological samples harvested perioperatively and during follow-up, and to correlate results with clinical end points.
Time Frame: 20 years
Reporting Status: Not Posted

10. Secondary Outcome: Anti-tumor Immunology
Description: The aim is to evaluate immunological parameters related to anti-tumor immunity and inflammatory factors
Time Frame: 20 years
Reporting Status: Not Posted

11. Secondary Outcome: Imaging
Description: The aim is to evaluate two new imaging methods, CT perfusion of liver and LIME-PET, in order to optimize the preoperative identification of colorectal liver metastases.
Time Frame: 5 years
Reporting Status: Not Posted

12. Secondary Outcome: Severity of Morbidity
Description: Severity of complications will be assessed by the Comprehensive Complication Index and the Accordion system
Time Frame: 30 days
Reporting Status: Not Posted

13. Secondary Outcome: Level of Adhesions
Description: Level of adhesions will be recorded during repeated liver resection in patients formerly randomized to open or laparoscopic liver resection. a modified version of the peritoneal adhesion index will be used for scoring.
Time Frame: 2 years
Reporting Status: Not Posted

14. Secondary Outcome: Number of Patients That Complete Adjuvant Oncologic Treatment
Description: Time from operation to initiation of oncologic treatment, and the total number of courses given will be recorded and compared between the groups.
Time Frame: 1 year
Reporting Status: Not Posted

15. Secondary Outcome: Readmissions
Description: Readmissions within 30 days after surgery will be recorded, both admissions to Oslo University Hospital and to referring hospitals.
Time Frame: 30 days
Reporting Status: Not Posted

16. Secondary Outcome: Incidence of Incisional Hernia
Description: CT scans will be performed to examine for incisional hernia 1 year after surgery
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were systematically collected using the Accordion system
Arm/Group | Open Liver Resection | Laparoscopic Liver Resection
All-Cause Mortality (participants affected / at risk) | 1/147 | 0/133
Serious Adverse Events (participants affected / at risk) | 10/147 | 4/133
Other Adverse Events (participants affected / at risk) | 0/147 | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Liver Resection (N=147) | Laparoscopic Liver Resection (N=133)
Bleeding (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Suspected bowel perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Fascia dehiscence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Small bowel perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Sudden death (General disorders) | 1 (1) | 0 (0)
Intraabdominal abcess (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes